CLINICAL TRIAL: NCT02203968
Title: Fibrinogen in the Initial Resuscitation of Severe Trauma (FiiRST): a Randomized Feasibility Trial
Brief Title: Fibrinogen in the Initial Resuscitation of Severe Trauma (FiiRST)
Acronym: FiiRST
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 064-2014
Record Dates: First submitted 2014-07-08; First posted 2014-07-30 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Trauma; Injury; Bleeding; Haemorrhage; Coagulopathy
Keywords: Fibrinogen replacement; Trauma coagulopathy; Hypofibrinogenemia; Early trauma coagulopathy; Haemorrhage; Fibrinogen concentrate; Feasibility trial; Clinical trials
MeSH Terms: conditions — Wounds and Injuries; Hemorrhage; Hemostatic Disorders; Afibrinogenemia | interventions — Fibrinogen; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Normal saline (Placebo Comparator): Placebo (normal saline) will be administered intravenously as a single 300ml rapid infusion (less than 3min) via level I automated pressure pump within one hour of hospital admission.
  Interventions: Drug: Placebo Comparator
- Fibrinogen concentrate (Active Comparator): Fibrinogen concentrate (RiaSTAP™) is a freeze-dried lyophilised plasma product presented in powdered form. The powder is reconstituted with water for intravenous injection at a concentration of 20 mg fibrinogen per ml. The concentrate is formulated with human albumin, L-arginine, sodium citrate and sodium chloride. RiaSTAP™ is supplied as a purified lyophilisate in a 1g dosage form and is reconstituted in 50 ml of sterile water. The final volume of RiaSTAP™ to be infused in this study will therefore be 300 ml.
  Interventions: Drug: Fibrinogen concentrate

INTERVENTIONS:
Drug: Fibrinogen concentrate — Six grams of fibrinogen concentrate (RiaSTAP™) will be administered intravenously as a single 300ml rapid infusion (less than 3min) via level I automated pressure pump within one hour of hospital admission.
  Other Names: RiaSTAP™
  Arms: Fibrinogen concentrate
Drug: Placebo Comparator — Placebo Comparator: Normal saline Placebo (normal saline) will be administered intravenously as a single 300ml rapid infusion (less than 3min) via level I automated pressure pump within one hour of hospital admission.
  Other Names: Normal saline
  Arms: Normal saline

SUMMARY:
Trauma is the leading cause of death in people 44 years of age or younger. After major trauma, such as following high-speed motor vehicle collision, bleeding coupled with clotting defects is responsible for most of deaths in the first hours of hospital admission. Of note, these bleeding-related deaths are potentially preventable. Accordingly, the initial in-hospital management of severely injured patients focuses on stopping bleeding, replacing blood loss and correcting clotting defects.

Recently, animal and human research demonstrated that one of the major clotting defects following injury and bleeding is the drop in blood levels of fibrinogen (a clotting factor), which is detected on hospital admission in severely injured patients. These low fibrinogen levels are associated with increased blood transfusion and death. However, in North America, the standard of care for replacing low fibrinogen requires the use of cryoprecipitate, which is a frozen blood product with long preparation time, and similarly to other blood products, carries the risk of viral transmission and transfusion complications. Alternately, many Europeans countries where cryoprecipitate has been withdrawn from the market due to safety concerns, use fibrinogen concentrate. Fibrinogen concentrate undergoes pathogen inactivation, which is a process to eliminate the risk of transmitting viruses, bacteria and parasites, is likely a safer and faster alternative to cryoprecipitate. In Canada, fibrinogen concentrate is licensed for congenital low fibrinogen only.

Although preliminary data suggest that fibrinogen supplementation in trauma is associated with reduced bleeding, blood transfusion, and death, the feasibility, safety and efficacy of early fibrinogen replacement remains unknown. We proposed to conduct a feasibility randomized trial to evaluate the use of early fibrinogen concentrate against placebo in injured patients at our trauma centre.

A pilot trial is necessary to demonstrate the feasibility of rapidly preparing, delivering, and infusing fibrinogen concentrate as an early therapy to prevent excessive bleeding in trauma. This feasibility trial will provide preliminary safety and clinical outcome data to inform the design of larger trials; which ultimately aims to prevent bleeding-related deaths in the trauma population.

ELIGIBILITY:
Inclusion Criteria:

1. Injured trauma (penetrating or blunt) patients who are at risk of significant bleeding, defined as: i. Systolic blood pressure (SBP) ≤ 100mmHg at any time from the injury scene until 30min after hospital admission AND ii. Red blood cell transfusion has been ordered by the trauma team leader (or delegate)

Exclusion Criteria:

1. Patients in shock which the etiology is purely not related to bleeding:

   i. Cardiogenic (myocardial or valvular dysfunction); ii. Distributive (septic, anaphylactic, acute adrenal insufficiency and neurogenic) and iii. Obstructive (cardiac tamponade, tension pneumothorax and massive pulmonary emboli).
2. Severe head injury, defined as any of the following:

   i. Glasgow coma scale (GCS) of 3 due to severe traumatic brain injury (TBI); ii. TBI with clear indication of immediate neurosurgical intervention based on clinical findings (mechanism of trauma associated with focal signs such as anisocoria with fixed pupil) or on CT results (bleeding causing mass effect); iii. Unsalvageable head injury such as through-through gunshot wound to the head, open skull fracture with exposure/loss of brain tissue; as per the trauma team or neurosurgery initial clinical assessment or as per initial CT of the head findings;
3. Known complete or incomplete spinal cord injury;
4. Known hereditary or acquired coagulopathies unrelated to the trauma resuscitation (e.g. known hepatic dysfunction);
5. Use of anticoagulant medications such as warfarin, low-molecular weight heparin, and direct thrombin and factor Xa inhibitors;
6. Moribund with evidence of unsalvageable injuries and withdrawal of care, as per the trauma team;
7. Received blood products prior to admission;
8. Patients with estimated body weight under 50Kg;
9. Patients with known or suspected pregnancy;
10. Patients arriving more than 6hr after injury.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Feasibility | One year
  1.Feasibility endpoint: 1.1Proportion of patients receiving study intervention (Fibrinogen Concentrate [FC] or placebo) within first hour of hospital admission. Based on the trial's sample size of 50 patients, feasibility is defined by 85% (96% confidence interval (CI) [72% - 98%]) of study participants receiving the study intervention within the first hour of hospital admission

SECONDARY OUTCOMES:
Other feasibility endpoints and physiologic endpoints | one year
  Other feasibility endpoints:1.2.Proportion of patients receiving study intervention prior to any blood transfusion; 1.3.Times to randomization, issue, and start of infusion; 1.4.Duration of infusion; 1.5.Wastage of study intervention; 1.6.Proportion of patients with blood tests performed for all time points; 1.7.Proportion of missed patients (eligible but not randomized); 1.8.Randomization errors.
  Physiologic endpoints: Plasma fibrinogen levels; Rotational Thromboelastometry/ Thromboelastography parameters (functional fibrinogen, fibtem, fibtem plus); plasmin anti-plasmin complex; tissue plasminogen activator; plasminogen activator inhibitor-1; d-dimer levels; international normalized ratio [INR]; partial thromboplastin time; complete blood count; endogenous thrombin potential; factor XIII; factor V; and activated protein C will be obtained on admission; and +1h, +3h, +11h, +23h & +47h following start time of study infusion

OTHER OUTCOMES:
Clinical Parameters | one year
  Rates of symptomatic thromboembolic complications in both study arms defined by the evidence of any of the following any time during hospital stay: deep venous thrombosis; myocardium infarction; cerebral vascular accident; pulmonary embolism; and arterial thrombosis
  Rates of asymptomatic deep venous thrombosis by leg doppler at day 7 of hospital stay
  Mortality by exsanguination
  All-cause mortality at 28 days (mainly due to exsanguination; mainly neurological/ due to traumatic brain injury/ withdrawal of care; or mainly due to multiple organ failure/sepsis)
  Incidence of acute lung injury/ acute respiratory distress syndrome before day 28
  Multiple organ failure
  Total amount of crystalloids used in 24h
  Units of blood and blood products transfused in 24h of hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Barto Nascimento, MD MSc, Principal Investigator — Sunnybrook Health Sciences Centre, University of Toronto
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada